CLINICAL TRIAL: NCT03646539
Title: Randomized Clinical Trial of an Automated Conversational Agent Versus Treatment as Usual for the Management of Perinatal Mood
Brief Title: RCT of Automated Conversational Agent vs. Treatment as Usual for the Management of Perinatal Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amy Judy, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-46467
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Cognitive Therapy; Depression, Postpartum; Mental Health; Depression; Depressive Disorder; Anxiety; Telemedicine
Keywords: Automated conversational agent
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being; Depression; Depressive Disorder; Anxiety Disorders | interventions — Amyloid; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone use + treatment as usual (Experimental): Participants will receive treatment as usual and use the smartphone app for the management of mood.
  Interventions: Behavioral: Use of smartphone application (app); Other: Treatment as usual
- Treatment as usual (Active Comparator): Participants will receive treatment as usual.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Use of smartphone application (app) — Use of a CBT-based automated conversational agent available as a mobile device smartphone application for the management of mood.
  Arms: Smartphone use + treatment as usual
Other: Treatment as usual — Treatment as usual will include (but may not be limited to) the participant's 6-week postpartum follow-up visit with their obstetrics care team. Participants will be sent surveys to evaluate their depressive and anxiety symptoms.

SUMMARY:
The purpose of this study is to investigate the efficacy of an evidence-based smartphone application (app) for the management of mood compared to treatment as usual alone among 135 women who have been discharged post-delivery from Labor and Delivery at Stanford Children's Health - Lucile Packard Children's Hospital. Using psychometrically validated surveys for depression, postpartum depression, and anxiety, this study will evaluate whether the smartphone app has a differential effect on the mental health of postpartum women as compared to treatment as usual.

DETAILED DESCRIPTION:
The intervention is a cognitive behavioral therapy (CBT) based automated conversational agent available as a mobile device smartphone application. When a user logs in with the app, it asks questions about that user, such as how they're feeling, and the user is able to type their response, similar to texting or messaging. The app is then available for use by the user anytime (24 hours per day 7 days per week), and will check in with the user to encourage mood tracking followed by tailored delivery of CBT-based tools and other general psychoeducation. This smartphone app interacts with conversational tones, and offers empathy and behavioral pattern insight to users. The app's artificial intelligence becomes more specific to a user over time, based on conversations. The app allows patients are able to immediately process and receive empathy for significant events and removes barriers traditionally limiting treatment access (cost, stigma, health care system navigability, and lack of childcare or transportation).

ELIGIBILITY:
Inclusion Criteria:

* Postpartum day 0-7 after delivery
* Medically stable and cleared for discharge
* Owns smartphone
* English-speaking (because all intervention materials are in English)

Exclusion Criteria:

* Neonatal demise this admission
* Intrauterine fetal demise this admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in Patient Health Questionnaire (PHQ-9) scores at 6 weeks post-delivery | Baseline; 6 weeks post-delivery
  PHQ-9 will be used to assess depression. The maximum score is 27. The scale is interpreted as follows: 0-4 no depression, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Mean change from baseline in Edinburgh Postnatal Depression Scale Scores at 6 weeks | Baseline; 6 weeks post-delivery
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report used to measure postpartum depression (range 0-30, higher score indicates greater symptom burden). A score of >9 is indicative of perinatal major depression.

SECONDARY OUTCOMES:
Mean change from baseline in Patient Health Questionnaire (PHQ-9) scores at 2 weeks post-delivery | Baseline; 2 weeks post-delivery
  PHQ-9 will be used to assess depression. The maximum score is 27. The scale is interpreted as follows: 0-4 no depression, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Mean change from baseline in Patient Health Questionnaire (PHQ-9) scores at 4 weeks post-delivery | Baseline; 4 weeks post-delivery
  PHQ-9 will be used to assess depression. The maximum score is 27. The scale is interpreted as follows: 0-4 no depression, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Mean change from baseline in Edinburgh Postnatal Depression Scale Scores at 2 weeks | Baseline; 2 weeks post-delivery
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report used to measure postpartum depression (range 0-30, higher score indicates greater symptom burden). A score of >9 is indicative of perinatal major depression.
Mean change from baseline in Edinburgh Postnatal Depression Scale Scores at 4 weeks | Baseline; 4 weeks post-delivery
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report used to measure postpartum depression (range 0-30, higher score indicates greater symptom burden). A score of >9 is indicative of perinatal major depression.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Judy, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Department of Obstetrics and Gynecology, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005